CLINICAL TRIAL: NCT03172611
Title: A Defined, Plant-based, 4-week Dietary Intervention Reduces Lp(a) and Other Atherogenic Particles
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Texas Woman's University (Other)
Collaborators: Montgomery Heart & Wellness (Unknown)
Responsible Party: Principal Investigator, Rami Najjar, Principal Investigator, Texas Woman's University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 192790
Record Dates: First submitted 2017-05-29; First posted 2017-06-01 (Actual); Last update posted 2017-06-01 (Actual); Status verified 2017-05

CONDITIONS: Hypercholesterolemia
MeSH Terms: conditions — Hypercholesterolemia | interventions — Diet Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Plant-based diet (Experimental): A defined, plant-based diet was prescribed for 4 weeks.
  Interventions: Other: Dietary Intervention

INTERVENTIONS:
Other: Dietary Intervention — Subjects consumed a defined, plant-based diet for 4-weeks. Emphasized were raw fruits and vegetables.

SUMMARY:
This study evaluates the effects of consuming a defined, plant-based diet on lipoprotein(a) and other atherogenic particles associated with cardiovascular disease risk.

DETAILED DESCRIPTION:
Lipoprotein(a) is a carrier of oxidized low-density lipoprotein and is a particularly atherogenic biomarker. Lp(a) has been previously documented to be resistant to dietary therapies and its concentration is thought to be determined by genes. A plant-based diet has not been previously used in an attempt to influence the concentration of Lp(a).

Participants were instructed to follow a defined, plant-based dietary intervention for four weeks. All animal products were excluded. Cooked foods, free oils, soda, alcohol, and coffee were also to be excluded. All meals and snacks were provided to the participants for the full duration of the intervention. Emphasized were raw fruits and vegetables, while seeds, avocado, raw oats, raw buckwheat, and dehydrated foods were prepared as condiments. Vitamin, herbal, and mineral supplements were to be discontinued unless otherwise clinically indicated. Participants were not advised to alter their exercise habits.

Serum biomarkers were obtained from participants at baseline and after 4-weeks.

ELIGIBILITY:
Inclusion Criteria:

* Body Mass Index ≥25.0 kg/m^2
* Serum low-density lipoprotein cholesterol concentration ≥100
* Systolic blood pressure ≥140 mmHg or diastolic blood pressure ≥90

Exclusion Criteria:

* Tobacco use
* Drug abuse
* Excessive alcohol consumption (>2 glasses of wine or alcohol equivalent per day for men or >1 glass of wine or alcohol equivalent for woman)
* Current cancer diagnosis
* Estimated glomerular filtration rate <60 mg/dL
* Clinically defined infection
* Mental disability
* Hospitalization <6 months
* Previous exposure to plant-based diet

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 33 (Actual)
Dates: Start 2017-01-03 (Actual); Primary Completion 2017-03-08 (Actual); Study Completion 2017-03-15 (Actual)

PRIMARY OUTCOMES:
Change in serum lipoprotein(a) | Baseline and 4-weeks
  Serum Lp(a) (nmol/L) was documented at baseline and after 4-weeks

SECONDARY OUTCOMES:
Change in serum total cholesterol | Baseline and 4-weeks
  Serum total cholesterol (mg/dL) was documented at baseline and after 4-weeks
Change in serum low-density lipoprotein cholesterol | Baseline and 4-weeks
  LDL cholesterol (mg/dL) was documented at baseline and after 4-weeks
Change in serum high-density lipoprotein cholesterol | Baseline and 4-weeks
  Serum HDL (mg/dL) was documented at baseline and after 4-weeks
Change in serum apolipoprotein-B | Baseline and 4-weeks
  Serum Apo-B (mg/dL) was documented at baseline and after 4-weeks
Change in serum low-density lipoprotein particles | Baseline and 4-weeks
  Serum LDL-P (nmol/L) was documented at baseline and after 4-weeks
Change in serum small-dense low-density lipoprotein cholesterol | Baseline and 4-weeks
  Serum sdLDL-C (mg/dL) was documented at baseline and after 4-weeks
Change in serum high-density lipoprotein 2 cholesterol | Baseline and 4-weeks
  Serum HDL2-C (mg/dL) was documented at baseline and after 4-weeks
Change in serum apolipoprotein A-1 | Baseline and 4-weeks
  Serum Apo A-1 (mg/dL) was documented at baseline and after 4-weeks

CONTACTS AND LOCATIONS:
Overall Officials: Rami Najjar, M.S., Principal Investigator — Texas Woman's University
Locations (1):
- Montgomery Heart & Wellness, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Brown SA, Morrisett J, Patsch JR, Reeves R, Gotto AM Jr, Patsch W. Influence of short term dietary cholesterol and fat on human plasma Lp[a] and LDL levels. J Lipid Res. 1991 Aug;32(8):1281-9. PMID 1837559
- [Background] Bloomer RJ, Kabir MM, Canale RE, Trepanowski JF, Marshall KE, Farney TM, Hammond KG. Effect of a 21 day Daniel Fast on metabolic and cardiovascular disease risk factors in men and women. Lipids Health Dis. 2010 Sep 3;9:94. doi: 10.1186/1476-511X-9-94. PMID 20815907
- [Background] Jenkins DJ, Kendall CW, Popovich DG, Vidgen E, Mehling CC, Vuksan V, Ransom TP, Rao AV, Rosenberg-Zand R, Tariq N, Corey P, Jones PJ, Raeini M, Story JA, Furumoto EJ, Illingworth DR, Pappu AS, Connelly PW. Effect of a very-high-fiber vegetable, fruit, and nut diet on serum lipids and colonic function. Metabolism. 2001 Apr;50(4):494-503. doi: 10.1053/meta.2001.21037. PMID 11288049
- [Background] Le LT, Sabate J. Beyond meatless, the health effects of vegan diets: findings from the Adventist cohorts. Nutrients. 2014 May 27;6(6):2131-47. doi: 10.3390/nu6062131. PMID 24871675
- [Background] Jenkins DJ, Kendall CW, Marchie A, Parker TL, Connelly PW, Qian W, Haight JS, Faulkner D, Vidgen E, Lapsley KG, Spiller GA. Dose response of almonds on coronary heart disease risk factors: blood lipids, oxidized low-density lipoproteins, lipoprotein(a), homocysteine, and pulmonary nitric oxide: a randomized, controlled, crossover trial. Circulation. 2002 Sep 10;106(11):1327-32. doi: 10.1161/01.cir.0000028421.91733.20. PMID 12221048
- [Background] Kiortsis DN, Tzotzas T, Giral P, Bruckert E, Beucler I, Valsamides S, Turpin G. Changes in lipoprotein(a) levels and hormonal correlations during a weight reduction program. Nutr Metab Cardiovasc Dis. 2001 Jun;11(3):153-7. PMID 11590990